CLINICAL TRIAL: NCT05819619
Title: Prophylactic Analgesic and Antiemetic Regimen for Medical Abortion < 70 Days
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Inability to recruit and staffing changes
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2021-1405
Record Dates: First submitted 2023-03-15; First posted 2023-04-19 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Nausea; Pain
Keywords: medical abortion; prophylactic use; nausea; pain; patient satisfaction
MeSH Terms: conditions — Nausea; Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Administration of ibuprofen or ondansetron only when experiencing pain or nausea respectively post misoprostol administration.
  Interventions: Drug: Use of ibuprofen and ondansetron at symptom onset post misoprostol administration
- Prophylactic use (Experimental): Administration of ibuprofen and ondansetron at the time of misoprostol administration.
  Interventions: Drug: Prophylactic use of ibuprofen and ondansetron post misoprostol administration

INTERVENTIONS:
Drug: Prophylactic use of ibuprofen and ondansetron post misoprostol administration — Prophylactic use of ibuprofen and ondansetron post misoprostol administration
  Arms: Prophylactic use
Drug: Use of ibuprofen and ondansetron at symptom onset post misoprostol administration — Administration of ibuprofen or ondansetron only when experiencing pain or nausea respectively post misoprostol administration.
  Arms: Standard of care

SUMMARY:
Randomized trial which will aim to evaluate whether prophylactic use of ondansetron and ibuprofen will decrease side effects associated with medical abortion and increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* English speaking
* female volunteers undergoing medical abortion whether for voluntary interruption of pregnancy or missed abortion
* Gestational age </= 70 days confirmed via ultrasound
* Access to a time keeping device
* Willingness to complete a telephone or in-clinic follow up

Exclusion Criteria:

* chronic medical problems including but not limited to cardiac conditions, malignancy or organ damage
* Failed medical abortion resulting in surgical management
* Known intrauterine infection
* Known allergy to ondansetron or ibuprofen
* Subjects chronically receiving analgesic drugs
* Subjects unable to give consent
* Subjects taking medications that interact with ondansetron or ibuprofen

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Figueroa, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Antonia Oladipo, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Prophylactic Use
Started | 3 | 5
Completed | 0 | 3
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Prophylactic Use | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 29 [21 to 41] | 29 [22 to 38] | 29 [21 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 1 | 1 | 2
  Non Hispanic/Latino | 1 | 2 | 3
  Other- Hispanic/Latino Hispanic/Latino | 0 | 1 | 1
  Central or South American | 0 | 1 | 1
  Cuban | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Determine if prophylactic use of ondansetron and ibuprofen during medical abortion treatment can increase patient satisfaction thereby creating a more favorable outcome.
  Patient satisfaction will be assessed using a home developed survey. Satisfaction is measured on 5-Likert scale ranging from Very satisfied to Very dissatisfied.
Time Frame: At follow up visit, within 2 weeks from the administration of misoprostol
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 4
Participants
  Very satisfied | 1 | 1
  Fairly satisfied | 2 | 2
  Neither satisfied nor dissatisfied | 0 | 1

2. Primary Outcome: Patient Satisfaction Based on Recommendation of Regimen
Description: Determine if prophylactic use of ondansetron and ibuprofen during medical abortion treatment can increase patient satisfaction based on their likelihood to recommend the regimen.
  Likelihood to recommend will be assessed using a home developed survey measured on 5-Likert scale ranging from "Extremely likely to recommend" to "Extremely unlikely to recommend" (an additional "I do not know option" will be provided).
Time Frame: At follow up visit, within 2 weeks from the administration of misoprostol
Population: Patients who were part of the active cohort and got the prophylactic administration
Measure: Count of Participants; unit: Participants
Groups:
- Prophylactic Group: Administration of ibuprofen and ondansetron at the time of misoprostol administration.
  Prophylactic use of ibuprofen and ondansetron post misoprostol administration: Prophylactic use of ibuprofen and ondansetron post misoprostol administration
Arm/Group | Prophylactic Group
Number analyzed (Participants) | 4
Participants
  Extremely likely to recommend | 1
  Likely to recommend | 2
  Neither likely nor unlikely to recommend | 1
  Unlikely to recommend | 0
  Extremely unlikely to recommend | 0
  I do not know | 0

3. Secondary Outcome: Pain Management at 6-8 Hours
Description: Evaluate for a satisfactory pain management regimen for medical abortion using a numerical pain scale ranging from 1 to 10 with 1 being "no pain" and 10 being "very much pain".
Time Frame: Within 6-8 hours from the administration of misoprostol
Measure: Mean (Full Range); unit: score on a pain scale
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 4
score on a pain scale | 7.66 [7 to 10] | 6.5 [3 to 9]

4. Secondary Outcome: Pain Management at 24 Hours
Description: as for outcome 3
Time Frame: Within 24 hours from the administration of misoprostol
Measure: Mean (Full Range); unit: score on a pain scale
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 4
score on a pain scale | 5 [2 to 8] | 4.8 [1 to 9]

5. Secondary Outcome: Nausea Management
Description: Evaluate for a satisfactory anti-nausea management regimen for medical abortion using a numerical nausea scale ranging from 1 to 10 with 1 being "no nausea" and 10 being "very much nausea".
Time Frame: Within 6-8 hours from the administration of misoprostol
Measure: Mean (Full Range); unit: score on a nausea scale
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 4
score on a nausea scale | 4.33 [1 to 8] | 4 [1 to 7]

6. Secondary Outcome: Nausea Management
Description: as for outcome 5
Time Frame: Within 24 hours from the administration of misoprostol
Measure: Mean (Full Range); unit: score on a nausea scale
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 5
score on a nausea scale | 3 [1 to 7] | 1.2 [1 to 2]

7. Secondary Outcome: Need for Pain Management Medication.
Description: Evaluate for a satisfactory pain management regimen for medical abortion based on the need for additional pain medication (Yes vs. No).
Time Frame: Within 24 hours from the administration of misoprostol
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 5
Participants
  Yes | 3 | 2
  No | 0 | 3

8. Secondary Outcome: Need for Anti-nausea Medication.
Description: Evaluate for a satisfactory anti-nausea management regimen for medical abortion based on the additional anti-nausea medication (Yes vs. No).
Time Frame: Within 24 hours from the administration of misoprostol
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Prophylactic Use
Number analyzed (Participants) | 3 | 5
Participants
  Yes | 1 | 0
  No | 2 | 5

ADVERSE EVENTS:
Time Frame: 24-hour follow-up
Arm/Group | Standard of Care | Prophylactic Use
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT05819619/Prot_SAP_000.pdf